CLINICAL TRIAL: NCT00094835
Title: An Open-label, Dose-finding Study to Evaluate the Safety and Pharmacokinetics (PK) of AMG 706 With Carboplatin/Paclitaxel, AMG 706 With Panitumumab and AMG 706 With Panitumumab and Carboplatin/Paclitaxel in the Treatment of Subjects With Advanced Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Study to Evaluate Motesanib With or Without Carboplatin/Paclitaxel or Panitumumab in the Treatment of Patients With Advanced Non-Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20040153; NCT00107224 (obsolete NCT alias)
Record Dates: First submitted 2004-10-27; First posted 2004-10-27 (Estimated); Results first posted 2014-03-24 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-02

CONDITIONS: Lung Cancer; Non-Small Cell Lung Cancer
Keywords: Lung cancer, Non-small cell lung cancer, NSCLC; Clinical Trial, Panitumumab, AMG 706; Anti-angiogenesis; Immunex, Abgenix, Amgen; Stage IIIB, Stage IV, Unresectable
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — Panitumumab; motesanib diphosphate; Paclitaxel; Carboplatin

ARMS (3):
- Paclitaxel + Carboplatin + Motesanib (Experimental): Chemotherapy naïve participants received paclitaxel 200 mg/m^2 and carboplatin chemotherapy administered by intravenous (IV) infusion on Day 1 of each 21-day cycle, and motesanib, orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter. The initial dose of motesanib was 50 mg once daily administered in the initial cohort and up to 125 mg once daily was used in subsequent cohorts. A cycle was defined as the 3 weeks plus the time to recover from toxicity, if encountered.
  Interventions: Drug: Motesanib diphosphate; Drug: Paclitaxel; Drug: Carboplatin
- Panitumumab + Motesanib (Experimental): Participants with no more than one prior chemotherapy regimen for NSCLC received panitumumab administered by IV at 9.0 mg/kg on Day 1 of each 21-day cycle, and motesanib, orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter. The initial dose of motesanib was 50 mg once daily administered in the initial cohort, up to 125 mg once daily was used in subsequent cohorts.
  Interventions: Biological: Panitumumab; Drug: Motesanib diphosphate
- Panitumumab + Paclitaxel + Carboplatin + Motesanib (Experimental): Chemotherapy naïve participants received panitumumab administered by IV at 9.0 mg/kg on Day 1 of each 21-day cycle, paclitaxel 200 mg/m^2 and carboplatin chemotherapy administered by IV infusion on Day 1 of each 21-day cycle, and motesanib, orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter.
  Participants were enrolled in this arm once a safe and tolerable dose of motesanib was established.
  Interventions: Biological: Panitumumab; Drug: Motesanib diphosphate; Drug: Paclitaxel; Drug: Carboplatin

INTERVENTIONS:
Biological: Panitumumab — 9.0 mg/kg on Day 1 of each 21-day cycle administered by intravenous infusion over approximately 60 minutes.
  Other Names: Vectibix; ABX-EGF
  Arms: Panitumumab + Motesanib; Panitumumab + Paclitaxel + Carboplatin + Motesanib
Drug: Motesanib diphosphate — Dose-finding with an initial dose of 50 mg once daily and up to 125 mg once daily. 75 mg twice daily was also to be tested.
  Other Names: AMG 706
Drug: Paclitaxel — Paclitaxel 200 mg/m^2 administered by IV infusion over 3 hours.
  Arms: Paclitaxel + Carboplatin + Motesanib; Panitumumab + Paclitaxel + Carboplatin + Motesanib
Drug: Carboplatin — Carboplatin was administered IV over approximately 30 minutes. Carboplatin was dosed using the glomerular filtration rate (GFR) and Calvert formula to AUC/time curve of 6 mg/mL×min.
  Arms: Paclitaxel + Carboplatin + Motesanib; Panitumumab + Paclitaxel + Carboplatin + Motesanib

SUMMARY:
The purpose of this trial is: - To characterize the safety profile of motesanib when used in combination with carboplatin/paclitaxel (CP), with panitumumab or with CP and panitumumab in patients with advanced non-small cell lung cancer (NSCLC). - To establish the pharmacokinetic (PK) profile of motesanib when it is used in combination with CP, with panitumumab, or with CP and panitumumab. - To compare the paclitaxel and motesanib PK profiles when the medications are administered 30 minutes (min) or approximately 48 hours (hrs) apart. - To characterize the panitumumab and paclitaxel exposure in the combination regimens of motesanib with CP, motesanib with panitumumab, or motesanib with CP and panitumumab. - To describe the objective response rate (ORR) in each dose cohort. - To measure the immunogenicity of panitumumab in patients administered motesanib with panitumumab and motesanib with CP and panitumumab.

DETAILED DESCRIPTION:
This was a multicenter, open-label, dose-finding clinical trial examining the safety and PK of once or twice daily motesanib administered with CP or with CP and panitumumab in chemotherapy naïve patients, and with panitumumab in patients with no more than one prior chemotherapy regimen for NSCLC.

Participants were enrolled into the Panitumumab + Paclitaxel + Carboplatin + Motesanib once a safe and tolerable dose of AMG 706 was established in the other treatment arms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of unresectable stage IIIB or IV non-small cell lung cancer (NSCLC)
* No more than one prior chemotherapy
* Adequate hematologic, renal and hepatic function
* Measurable disease or evaluable disease on CAT scan or MRI
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Able to fast for 10 hrs twice during the study - Able to tolerate oral medications
* Life expectancy of at least 3 months

Exclusion Criteria:

* Symptomatic or untreated central nervous system metastases requiring current treatment
* History of arterial thrombosis within 1 year prior to enrollment
* Anticoagulant therapy, except for warfarin of less than 2mg per day
* Symptomatic peripheral neuropathy
* History of pulmonary hemorrhage or hemoptysis
* Myocardial infarction within 1 year before enrollment
* Uncontrolled hypertension [diastolic greater than 85 mmHg; systolic greater than 145 mmHg]
* History of other cancer, unless treated with no known active disease for longer than 3 years
* Previous treatment with AMG 706 or panitumumab, previous treatment with inhibitors of VEGF or EGF
* No antibody treatment for 6 weeks prior to enrollment
* Known HIV positive, hepatitis C positive or hepatitis B surface antigen positive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2005-01; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Background] Blumenschein GR Jr, Reckamp K, Stephenson GJ, O'Rourke T, Gladish G, McGreivy J, Sun YN, Ye Y, Parson M, Sandler A. Phase 1b study of motesanib, an oral angiogenesis inhibitor, in combination with carboplatin/paclitaxel and/or panitumumab for the treatment of advanced non-small cell lung cancer. Clin Cancer Res. 2010 Jan 1;16(1):279-90. doi: 10.1158/1078-0432.CCR-09-1675. Epub 2009 Dec 22. PMID 20028752
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from 18 January 2005 through 25 September 2006
Groups:
- Paclitaxel/Carboplatin + Motesanib 50 mg QD: Chemotherapy naïve participants received paclitaxel 200 mg/m^2 and carboplatin chemotherapy administered by intravenous (IV) infusion on Day 1 of each 21-day cycle, and motesanib, 50 mg once daily (QD) orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter.
- Paclitaxel/Carboplatin + Motesanib 125 mg QD: Chemotherapy naïve participants received paclitaxel 200 mg/m^2 and carboplatin chemotherapy administered by intravenous (IV) infusion on Day 1 of each 21-day cycle, and motesanib, 125 mg QD orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter.
- Paclitaxel/Carboplatin + Motesanib 75 mg BID: Chemotherapy naïve participants received paclitaxel 200 mg/m^2 and carboplatin chemotherapy administered by intravenous (IV) infusion on Day 1 of each 21-day cycle, and motesanib, 75 mg twice daily (BID) orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter.
- Panitumumab + Motesanib 50 mg QD: Participants with no more than one prior chemotherapy regimen for NSCLC received panitumumab 9.0 mg/kg IV on Day 1 of each 21-day cycle, and motesanib 50 mg QD, orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter.
- Panitumumab + Motesanib 125 mg QD: Participants with no more than one prior chemotherapy regimen for NSCLC received panitumumab 9.0 mg/kg IV on Day 1 of each 21-day cycle, and motesanib 125 mg QD, orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter.
- Panitumumab + Motesanib 75 mg BID: Participants with no more than one prior chemotherapy regimen for NSCLC received panitumumab 9.0 mg/kg IV on Day 1 of each 21-day cycle, and motesanib 75 mg BID, orally self-administered on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter.
- Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD: Chemotherapy naïve participants received panitumumab 9.0 mg/kg, paclitaxel 200 mg/m^2 and carboplatin chemotherapy administered by IV infusion on Day 1 of each 21-day cycle, and motesanib 125 mg QD, orally on Days 3-21 of Cycle 1 and then on Days 1 to 21 of Cycle 2 and all cycles thereafter.
Period: Overall Study
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Started | 9 | 11 | 7 | 5 | 7 | 6 | 6
Treated With Motesanib | 6 | 11 | 6 | 4 | 7 | 5 | 6
Completed | 5 | 8 | 4 | 4 | 3 | 3 | 4
Not Completed | 4 | 3 | 3 | 1 | 4 | 3 | 2
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Non-compliance | 1 | 2 | 2 | 0 | 2 | 2 | 1
Not completed — Other | 1 | 1 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The analysis is based on the Safety Analysis Set which consists of all consented participants who received at least one dose of motesanib.
Groups:
- Total: Total of all reporting groups
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD | Total
Number analyzed (Participants) | 6 | 11 | 6 | 4 | 7 | 5 | 6 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (7.8) | 55.7 (12.7) | 64.5 (6.1) | 57.5 (9.9) | 64.0 (9.6) | 51.6 (14.6) | 59.0 (5.5) | 59.9 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 4 | 3 | 0 | 5 | 1 | 3 | 16
  Male | 6 | 7 | 3 | 4 | 2 | 4 | 3 | 29
Race/Ethnicity, Customized [Number; unit: participants]
  White or Caucasian | 6 | 11 | 5 | 4 | 6 | 4 | 5 | 41
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2
  Black or African American | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time to Maximum Plasma Concentration of Motesanib (Tmax) for Cycle 1
Description: The time after dosing that the maximal plasma concentration of motesanib was observed in Cycle 1. For the 75 mg BID cohorts, Tmax is reported for the first daily dose.
Time Frame: Cycle 1, Day 3 at predose, 15 and 30 minutes, and at 1, 2, 4, 6, 10 (QD cohorts only), and 24 hours post-dose.
Population: The pharmacokinetic (PK) population consisted of all consented patients who received motesanib and had evaluable pharmacokinetic data and did not have significant protocol deviations that affected the data or key-dosing information that was missing.
Measure: Median (Full Range); unit: hours
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Number analyzed (Participants) | 4 | 9 | 6 | 4 | 6 | 3 | 3
hours | 0.75 [0.5 to 2.0] | 1.0 [0.5 to 6.0] | 0.75 [0.25 to 1.00] | 1.5 [0.5 to 4.0] | 1.0 [0.5 to 1.0] | 0.58 [0.50 to 1.00] | 1.0 [1.0 to 4.0]

2. Secondary Outcome: Percentage of Participants With an Overall Objective Response
Description: Confirmed objective tumor response defined as a complete response (CR) or partial response (PR) using modified Response Evaluation Criteria in Solid Tumors (RECIST) version 1.0. Tumor response was evaluated by computed tomography (CT) scan or magnetic resonance imaging (MRI). Responding disease (CR or PR) was confirmed no less than 4 weeks after the criteria for response were first met. A complete response defined as the disappearance of all target lesions and all non-target lesions, no new lesions and normalization of tumor marker level. Partial response defined as either the disappearance of all target lesions and the persistence of one or more non-target lesion(s) or/and maintenance of tumor marker level above the normal limits, or, at least a 30% decrease in the sum of the longest diamer (LD) of target lesions, taking as reference the baseline sum LD and no new lesions and/or unequivocal progression of existing non-target lesions.
Time Frame: After 9 weeks of treatment (at the end of Cycle 3)
Population: Efficacy analysis set, composed of all enrolled participants who received at least one dose of motesanib in treatment arms 1-3 or at least one dose of motesanib with one dose of panitumumab in treatmnt arms 4-7.
Measure: Number; unit: Percentage of participants
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Number analyzed (Participants) | 6 | 11 | 6 | 4 | 7 | 5 | 6
Percentage of participants | 33 | 18 | 0 | 0 | 0 | 0 | 17

3. Primary Outcome: Maximum Observed Plasma Concentration of Motesanib (Cmax) in Cycle 1
Description: The maximal observed plasma concentration of motesanib after a single dose dose in Cycle 1. For the 75 mg BID cohorts, Cmax is reported for the first daily dose.
Time Frame: Cycle 1, Day 3 at predose, 15 and 30 min, and at 1, 2, 4, 6, 10 (QD cohorts only), and 24 hours post-dose.
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Number analyzed (Participants) | 4 | 9 | 6 | 4 | 6 | 3 | 3
ng/mL | 158 (55) | 525 (250) | 448 (112) | 328 (214) | 444 (130) | 198 (55) | 360 (243)

4. Primary Outcome: Estimated Terminal-phase Half-life (t1/2,z) of Motesanib in Cycle 1
Description: The terminal-phase elimination half-life (t1/2,z) of motesanib was calculated as ln(2)/λz. The terminal elimination rate constant (λz) was determined by linear regression of the natural logarithms of at least the last 3 measurable concentrations during the terminal phase. For the 75 mg BID cohorts, t1/2,z is reported for the first daily dose.
Time Frame: Cycle 1, Day 3 at predose, 15 and 30 min, and at 1, 2, 4, 6, 10 (QD cohorts only), and 24 hours postdose.
Population: PK Population. Participants with elevated motesanib concentrations at 24 hours were excluded from the calculations. Summary results are not presented for the Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD treatment group for which the sample size was smaller than 3.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID
Number analyzed (Participants) | 3 | 7 | 6 | 4 | 4 | 3
hours | 7.34 (2.07) | 5.33 (1.05) | 5.77 (1.45) | 6.47 (2.31) | 7.57 (2.60) | 8.28 (2.62)

5. Primary Outcome: Area Under the Plasma Concentration-time Curve for Motesanib in Cycle 1
Description: Area under the plasma concentration-time curve for motesanib in Cycle 1 calculated using the using the linear/log trapezoidal method. AUC from time zero to infinity (AUC0-inf) is reported for the 50 and 125 mg QD cohorts and AUC from time 0 to 24 hours post-dose (AUC0-24) is reported for the 75 mg BID cohort, where AUC0-24 is the sum of AUC0-12 for the first and second daily dose.
Time Frame: Cycle 1, Day 3 at predose, 15 and 30 minutes, and at 1, 2, 4, 6, 10 (QD cohorts only), and 24 hours post-dose.
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID
Number analyzed (Participants) | 3 | 7 | 5 | 4 | 4 | 3
μg*hr/mL | 0.971 (0.300) | 3.21 (1.12) | 2.91 (1.01) | 1.74 (0.63) | 3.23 (1.83) | 2.04 (1.06)

6. Primary Outcome: Trough Plasma Concentration at 24 Hours Post-dose (C24) for Motesanib in Cycle 1
Description: The trough plasma concentration for motesanib at 24 hours postdose in Cycle 1. For the 75 BID cohort, C24 is the observed concentration at 24 hours (ie, after the second daily dose).
Time Frame: Cycle 1, Day 3, 24 hours post-dose
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID
Number analyzed (Participants) | 3 | 9 | 5 | 4 | 4 | 3
ng/mL | 9.12 (4.17) | 26.5 (16.8) | 56.7 (27.4) | 14.0 (11.7) | 32.5 (21.5) | 56.8 (21.1)

7. Primary Outcome: Time to Maximum Plasma Concentration of Motesanib (Tmax) in Cycle 2
Description: The time after dosing that the maximal plasma concentration of motesanib was observed in Cycle 2. For the 75 mg BID cohorts, Tmax is reported for the first daily dose.
Time Frame: Cycle 2, Day 1 at predose, 15 and 30 min, and at 1, 2, 4, 6, 10 (QD cohorts only), and 24 hours post-dose.
Population: PK population
Measure: Median (Full Range); unit: hours
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Number analyzed (Participants) | 4 | 9 | 6 | 4 | 6 | 3 | 3
hours | 1.5 [1.0 to 2.0] | 1.0 [0.5 to 4.0] | 0.63 [0.25 to 4.0] | 1.0 [0.5 to 2.0] | 0.75 [0.25 to 2.0] | 1.0 [0.50 to 2.0] | 2.0 [0.5 to 2.0]

8. Primary Outcome: Maximum Observed Plasma Concentration of Motesanib (Cmax) in Cycle 2
Description: The maximal observed plasma concentration of motesanib in Cycle 2, after multiple doses. For the 75 mg BID cohorts, Cmax is reported for the first daily dose.
Time Frame: Cycle 2, Day 1 at predose, 15 and 30 min, and at 1, 2, 4, 6, 10 (QD cohorts only), and 24 hours post-dose.
Population: PK population
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Number analyzed (Participants) | 4 | 9 | 6 | 4 | 6 | 3 | 3
ng/mL | 148 (25) | 748 (701) | 390 (319) | 265 (190) | 672 (336) | 242 (153) | 651 (605)

9. Primary Outcome: Estimated Terminal-phase Half-life (t1/2,z) of Motesanib in Cycle 2
Description: as for outcome 4
Time Frame: Cycle 2, Day 1 at predose, 15 and 30 min, and at 1, 2, 4, 6, 10 (QD cohorts only), and 24 hours post-dose.
Population: PK Population. Participants with elevated motesanib concentrations at 24 hours were excluded from the calculations. Summary results are not presented for three treatment groups for which the sample size was smaller than 3.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD
Number analyzed (Participants) | 5 | 5 | 3 | 3
hours | 6.41 (2.08) | 6.36 (1.70) | 7.08 (0.35) | 4.90 (1.21)

10. Primary Outcome: Area Under the Plasma Concentration-time Curve From Time 0 to 24 Hours Post-dose for Motesanib in Cycle 2
Description: Area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC0-24) for motesanib in Cycle 2 calculated using the using the linear/log trapezoidal method. For the 75 mg BID cohort AUC0-24 is the sum of AUC0-12 for the first and second daily dose.
Time Frame: Cycle 2, Day 1 at predose, 15 and 30 minutes, and at 1, 2, 4, 6, 10 (QD cohorts only), and 24 hours post-dose.
Population: PK Population. Participants with elevated motesanib concentrations at 24 hours were excluded from the calculations. Summary results are not presented for two treatment groups for which the sample size was smaller than 3.
Measure: Mean (Standard Deviation); unit: μg*hr/mL
Arm/Group | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Number analyzed (Participants) | 5 | 5 | 3 | 5 | 3
μg*hr/mL | 4.50 (2.62) | 3.11 (2.38) | 1.26 (0.61) | 3.92 (2.65) | 3.16 (1.20)

11. Primary Outcome: Trough Plasma Concentration at 24 Hours Post-dose (C24) for Motesanib in Cycle 2
Description: The trough plasma concentration for motesanib at 24 hours postdose in Cycle 2. For the 75 BID cohort, C24 is the observed concentration at 24 hours (ie, after the second daily dose).
Time Frame: Cycle 2, Day 1, 24 hours post-dose
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Number analyzed (Participants) | 5 | 5 | 3 | 5 | 3
ng/mL | 43.4 (44.8) | 45.4 (35.9) | 10.4 (5.3) | 61.1 (72.6) | 45.1 (37.9)

ADVERSE EVENTS:
Time Frame: First dose through 30 days after last dose; maximum time on treatment was 322 days.
Description: The table of Other Adverse Events summarizes non-serious occurrences of adverse events that exceeded a 5% frequency in any treatment arm.
Arm/Group | Paclitaxel/Carboplatin + Motesanib 50 mg QD | Paclitaxel/Carboplatin + Motesanib 125 mg QD | Paclitaxel/Carboplatin + Motesanib 75 mg BID | Panitumumab + Motesanib 50 mg QD | Panitumumab + Motesanib 125 mg QD | Panitumumab + Motesanib 75 mg BID | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD
Serious Adverse Events (participants affected / at risk) | 5/6 | 2/11 | 3/6 | 0/4 | 1/7 | 4/5 | 2/6
Other Adverse Events (participants affected / at risk) | 6/6 | 11/11 | 6/6 | 4/4 | 7/7 | 5/5 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/Carboplatin + Motesanib 50 mg QD (N=6) | Paclitaxel/Carboplatin + Motesanib 125 mg QD (N=11) | Paclitaxel/Carboplatin + Motesanib 75 mg BID (N=6) | Panitumumab + Motesanib 50 mg QD (N=4) | Panitumumab + Motesanib 125 mg QD (N=7) | Panitumumab + Motesanib 75 mg BID (N=5) | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD (N=6)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paclitaxel/Carboplatin + Motesanib 50 mg QD (N=6) | Paclitaxel/Carboplatin + Motesanib 125 mg QD (N=11) | Paclitaxel/Carboplatin + Motesanib 75 mg BID (N=6) | Panitumumab + Motesanib 50 mg QD (N=4) | Panitumumab + Motesanib 125 mg QD (N=7) | Panitumumab + Motesanib 75 mg BID (N=5) | Panitumumab + Paclitaxel/Carboplatin + Motesanib 125 mg QD (N=6)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 0 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 2 | 1 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Conduction disorder (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 1
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Ear discomfort (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Change of bowel habit (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 2 | 1 | 0 | 2 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 6 | 0 | 5 | 3 | 5
Dyspepsia (Gastrointestinal disorders) | 2 | 3 | 1 | 0 | 1 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2
Gastrointestinal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gingival pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Gingival ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 4 | 6 | 5 | 1 | 3 | 2 | 4
Odynophagia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 3 | 2 | 0 | 3 | 1 | 4
Vomiting (Gastrointestinal disorders) | 4 | 4 | 5 | 0 | 1 | 4 | 1
Adverse drug reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Chills (General disorders) | 0 | 1 | 2 | 1 | 0 | 0 | 0
Early satiety (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 5 | 8 | 4 | 2 | 6 | 5 | 5
Hypothermia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Irritability (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mucosal inflammation (General disorders) | 0 | 2 | 1 | 0 | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 0 | 0 | 0 | 0 | 1 | 0
Oedema (General disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 2 | 0 | 0 | 3 | 1
Temperature intolerance (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Escherichia bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infected cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 0 | 0
Liver abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lymph gland infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Oral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 0 | 0 | 1 | 1 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 0 | 0 | 0 | 0
Staphylococcal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tooth infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 2 | 0 | 1
Incision site complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Breath sounds abnormal (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 4 | 2 | 1 | 2 | 2 | 2
White blood cell count decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1 | 4 | 2 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 2 | 0 | 2 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 4 | 3 | 0 | 0 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 5 | 5 | 2 | 3 | 4 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 3 | 3 | 0 | 2 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 6 | 1 | 0 | 4 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 4
Shoulder pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Balance disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Coordination abnormal (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 2 | 0 | 1 | 1 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 1 | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 1 | 4 | 3 | 0 | 2 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 2 | 1 | 0 | 1 | 1 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0
Mental impairment (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Neuropathy (Nervous system disorders) | 4 | 3 | 2 | 0 | 0 | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 1 | 2 | 1 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 3 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 2 | 1 | 1 | 0 | 1 | 1
Confusional state (Psychiatric disorders) | 1 | 1 | 1 | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Personality change (Psychiatric disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Bladder pain (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Incontinence (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Allergic cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 1 | 2 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 2 | 0 | 3 | 0 | 2
Dyspnoea exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 4 | 1 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 2 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 1 | 1 | 0
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 4 | 1 | 0 | 2 | 0 | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1 | 3 | 3 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 2 | 2 | 0 | 1
Exfoliative rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 3 | 3 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 6 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0 | 0 | 2 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0
Rash follicular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 4 | 5 | 4 | 1 | 4 | 3 | 3
Hypotension (Vascular disorders) | 3 | 3 | 2 | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0
Thrombosis (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.